CLINICAL TRIAL: NCT03787108
Title: Measuring Fatty Liver With Ultrasound and MRS in Children With Overweight or Obesity (Dutch Title: Het Meten Van Leververvetting Met Echo en MRS in Kinderen Met Overgewicht of Obesitas)
Brief Title: Measuring Fatty Liver With Ultrasound and MRS in Children With Overweight or Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL64534.068.18
Record Dates: First submitted 2018-10-30; First posted 2018-12-26 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Fatty Liver Disease; Magnetic Resonance Spectroscopy; Ultrasonographic hepatorenal index
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with suspected NAFLD: Children with overweight or obesity. Both children that are and children that are not suspected of having NAFLD (based on ultrasound and laboratory findings) are included.
  Interventions: Other: Magnetic resonance spectroscopy measurement

INTERVENTIONS:
Other: Magnetic resonance spectroscopy measurement — Magnetic resonance spectroscopy measurement will be performed to measure liver fat content.

SUMMARY:
Obesity is associated with a variety of comorbidities, amongst which non-alcoholic fatty liver disease (NAFLD). A recent meta-analysis has shown that the prevalence of NAFLD in obese pediatric populations is around 35%, compared to approximately 8% in general pediatric populations, making it a very important health threat in these populations. The golden standard for diagnosis of NAFLD is liver biopsy. However, since liver biopsy is associated with a certain risk of morbidity and mortality, this method is inappropriate for screening large populations at-risk for developing NAFLD. Magnetic resonance spectroscopy has demonstrated excellent correlation with liver biopsy and the is the most accuratete non-invasive method to measure liver fat content in children. However, MRS is expensive and not available in all centres. A novel ultrasonographic measurement to quantitatively assess liver steatosis is the hepatorenal index (HRI). Previous studies have shown high sensitivity and specificity of the HRI, as compared to MRS and liver biopsy. However, this measurement has never been validated in children. In this study, the HRI will be compared to MRS in children with obesity, to validate the HRI and to determine cut-off points.

DETAILED DESCRIPTION:
Rationale: Obesity is associated with a variety of co-morbidities. Children with obesity are more likely to have risk factors associated with cardiovascular disease (eg, hypertension, high cholesterol, and type 2 diabetes mellitus), but also non-alcoholic fatty liver disease (NAFLD). A recent meta-analysis has shown that the prevalence of NAFLD in obese pediatric populations is approximately 35%, compared to approximately 8% in general pediatric populations [6], making it a very important health threat in these populations. The golden standard for the diagnosis of NAFLD is liver biopsy. However, since liver biopsy is associated with a certain risk of morbidity and mortality, this method is inappropriate for screening large populations at-risk for developing NAFLD. Magnetic resonance spectroscopy has demonstrated excellent correlation with liver biopsy and the most accurate non-invasive method to measure liver fat content in children. However, MRS is an expensive method that is not available in all centers. A novel ultrasonographic measurement to quantitatively assess liver steatosis is the hepatorenal index (HRI), which is calculated as the ratio of hepatic and renal ultrasonographic brightness. Previous studies in adults have shown a high sensitivity and specificity of the HRI, as compared to liver biopsy as well as H-MRS. However, the measurement of the HRI has never been validated in children. The validation of this simple, non-invasive method to quantitatively assess fat accumulation in the liver, could improve the screening for, and follow-up of, NAFLD in at-risk populations.

Objective: The aim of this study is to validate the ultrasonographic hepatorenal index in children with overweight, obesity and morbid obesity, by using MRS, and to determine cut-off points for the HRI according to liver fat percentages measured with MRS.

Study design: cross-sectional study

Study population: Overweight and obese children from the Centre for Overweight Adolescent and Childrens Healthcare (COACH) program.

Main study parameters/endpoints: Ultrasonographic hepato-renal index and liver fat percentage as determined by magnetic resonance spectroscopy.

Secondary study parameters/endpoints: correlate liver fat percentage as measured with MRS, and HRI, with anthropometric, metabolic and cardiovascular parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the COACH program
* Aged below 18 years

Exclusion Criteria:

* · Implanted medical devices such as pacemakers or neurostimulators

  * Metal objects in the body (for instances prosthetics, piercings, metal parts in the eye, permanent eyeliner)
  * Previous brain surgery
  * Cardiac arrhythmia
  * Epilepsy
  * Claustrofobia
  * Not wanting to be informed about accidental findings on MRS

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive participants in the COACH program (children with overweight or obesity), that meet the inclusion criteria, will be invited to participate in this study, until the calculated sample size is reached.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2019-03-31 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic hepato-renal index | Until december 2019
  Ratio of hepatic and renal echogenicity
Liver fat percentage | Until december 2019
  Liver fat percentage will be measured withmagnetic resonance spectroscopy.

SECONDARY OUTCOMES:
BMI z-score | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index
Liver enzyme levels | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index
Fibrosan values | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index
Lipid spectrum | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index
Glucose metabolism | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index
Blood pressure | Until december 2019
  Secondary outcomes will be correlated with liver fat percentage as measured with MRS and with the ultrasonographic hepato-renal index

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided